CLINICAL TRIAL: NCT04564794
Title: Prognostic Value of Low Irradiation Cardiac Stress Perfusion Scans
Brief Title: Prognostic Value of Cardial Stress Perfusion Imaging
Acronym: PROSPERCARS
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pierre Yves MARIE, Clinical director, Central Hospital, Nancy, France
Other Study IDs: 2020PI174
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
Keywords: coronary; myocardial perfusion tomoscintigraphy.
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stress myocardial perfusion scintigraphy is a reference examination for the detection and monitoring of coronary patients, and this examination has already been the subject of multiple validation studies, including for the stratification of the prognosis of these patients, information that can usefully guide therapeutic choices.

Today, this reduction in the activity of injected radiopharmaceuticals is taking place in a growing number of nuclear medicine departments.

The implications are unknown in terms of the risk of death of the different parameters studied

DETAILED DESCRIPTION:
Stress myocardial perfusion scintigraphy is a reference examination for the detection and monitoring of coronary patients, and this examination has already been the subject of multiple validation studies, including for the stratification of the prognosis of these patients, information that can usefully guide therapeutic choices (medical treatment, myocardial revascularization, ...). The arrival of new solid-state cameras has been a real technological leap for this examination, making it possible to significantly improve the quality of the images and also to drastically reduce the activities of injected radiopharmaceuticals and thus the exposure of patients and staff to ionizing radiation. Today, this reduction in the activity of injected radiopharmaceuticals is taking place in a growing number of nuclear medicine departments. The injected activities are reduced up to a third of those injected in the past (this is indeed the case in the population we propose to study).

However, the value of the prognostic stratification obtained with stress myocardial perfusion scans recorded with low activity on semiconductor cameras is not yet known. In particular, the implications are unknown in terms of the risk of death of the different parameters studied (normal or abnormal examination, extent of myocardial ischemia and infarction sequelae, impact on left ventricular function in post-stress and resting states, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Any coronary patient suspected or proven to have had a stress myocardial perfusion tomoscintigraphy performed at the Nancy CHRU and corresponding to a standardized model of expression of results (i.e. more than 10,000 reports).

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any coronary patient suspected or proven to have had a stress myocardial perfusion tomoscintigraphy performed at the Nancy CHRU and corresponding to a standardized model of expression of results (i.e. more than 10,000 reports).
Sampling Method: Probability Sample
Enrollment: 11952 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-11-26 (Actual)

PRIMARY OUTCOMES:
Overall mortality | 6 months
  to evaluate the prognostic contribution of low radiation stress myocardial perfusion scintigraphy on overall mortality risk , overall mortality will be calculate

SECONDARY OUTCOMES:
Death from cardiac causes, either proven or suspected (death from unexplained causes), | 6 months
  To evaluate the prognostic contribution of myocardial perfusion scintigraphy of low radiation stress on mortality from cardiac causes.
Major cardiac events (death of proven or suspected cardiac cause, myocardial infarction, myocardial revascularization procedure), | 6 months
  To evaluate the prognostic contribution of myocardial perfusion scintigraphy of low radiation stress on major cardiac events
Cardiac mortality and major cardiac events. | 6 months
  To evaluate the prognostic contribution of myocardial perfusion scintigraphy of low radiation stress on quality of examination complementary to coronary angiography in a subgroup of approximately 700 patients who had a coronary angiography within ≤ 2 months compared to scintigraphy.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Marie, MD, PhD, Study Director — Nancy CHRU hospital
Locations (1):
- Nancy Hospital, Vandœuvre-lès-Nancy, Grand Est, France

IPD SHARING:
Plan to Share IPD: No